CLINICAL TRIAL: NCT02665013
Title: Reducing Delay of Vaccination in Children Study
Acronym: REDIVAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: University of Colorado, Denver (Other); University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01HD079457-01 (NIH)
Record Dates: First submitted 2016-01-04; First posted 2016-01-27 (Estimated); Last update posted 2019-06-13 (Actual); Status verified 2019-04

CONDITIONS: Communicable Diseases
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tailored (Experimental): Participants will complete surveys at each intervention time point. Based on survey responses, they will receive vaccine information on the study website tailored to their vaccine concerns and values
  Interventions: Behavioral: Tailored
- Untailored (Placebo Comparator): Participants will complete surveys at each intervention time point and receive vaccine information on the study website. The vaccine information will NOT be tailored to their concerns and values.
  Interventions: Behavioral: Untailored
- Usual Care (No Intervention): Participants will complete surveys at each intervention time point. They will receive vaccine information sheets that are provided in the well child visits at enrollment in the study.

INTERVENTIONS:
Behavioral: Tailored — Pregnant women will be recruited to the study. The intervention will be delivered to participants prior to the child's 2 month well child visit, when the child is between 4 and 6 months of age, and when the child is 10-12 months of age. The first intervention occurs at enrollment in the study. Participants in the tailored intervention arm will receive vaccine information tailored specific to her concerns and values at each intervention point.
  Arms: Tailored
Behavioral: Untailored — Pregnant women will be recruited to the study. The intervention will be delivered to participants prior to the child's 2 month well child visit, when the child is between 4 and 6 months of age, and when the child is 10-12 months of age. The first intervention occurs at enrollment in the study. Participants in the untailored arm will receive vaccine information at each intervention time point, but it will not be tailored to her specific concerns.
  Arms: Untailored

SUMMARY:
This trial will assess the effectiveness of a tailored message intervention on decreasing infant undervaccination.

DETAILED DESCRIPTION:
This intervention is based on the concept of "message tailoring," whereby each mother is provided with individually customized vaccine- related information that addresses their unique concerns, values, questions and logistical barriers. Message tailoring is an evidence-based health messaging strategy that has been shown to improve compliance with a wide variety of preventive health care behaviors among diverse patient populations.

In this three-armed trial the investigator will examine how providing mothers with multiple "doses" of a tailored versus untailored version of our intervention compares with "usual care" for the impact on infant under-vaccination. Secondary outcomes will include maternal vaccine-related attitudes (including level of vaccine hesitancy), alignment of maternal values with provider recommendations, and self-efficacy for overcoming logistical barriers to vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled at Kaiser Permanente Colorado, Pregnant in the 3rd trimester, and plan to use Kaiser Permanente Colorado for the child's medical care received.

Exclusion Criteria:

* less then 18 years of age, non-english speaking and an inability to consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 824 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
The child's vaccination status | 200 days
  assessed using both a continuous and dichotomous measure. Continuous: measure of average days under-vaccinated is a recently developed metric measuring the average number of days a child is unvaccinated based on the vaccines given and the date when the vaccines where given. Dichotomous: mesauring the child's days undervaccinated or whether or not the child is up-to-date with no vaccination delays.

SECONDARY OUTCOMES:
Maternal Vaccine attitudes | 12 months
  Maternal vaccine attitudes are collected from survey items and include attitudes and beliefs about vaccines as well as level of vaccine hesitancy
Maternal Vaccine values | 12 months
  Health values related to vaccines are measured from survey items and include conformity, security, power, self-direction, and universalism

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Colorado, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Glanz JM, Wagner NM, Narwaney KJ, Pyrzanowski J, Kwan BM, Sevick C, Resnicow K, Dempsey AF. Web-Based Tailored Messaging to Increase Vaccination: A Randomized Clinical Trial. Pediatrics. 2020 Nov;146(5):e20200669. doi: 10.1542/peds.2020-0669. Epub 2020 Oct 12. PMID 33046584
- [Derived] Dempsey AF, Wagner N, Narwaney K, Pyrzanowski J, Kwan BM, Kraus C, Gleason K, Resnicow K, Sevick C, Cataldi J, Brewer SE, Glanz JM. 'Reducing Delays In Vaccination' (REDIVAC) trial: a protocol for a randomised controlled trial of a web-based, individually tailored, educational intervention to improve timeliness of infant vaccination. BMJ Open. 2019 May 22;9(5):e027968. doi: 10.1136/bmjopen-2018-027968. PMID 31122997

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT02665013/Prot_SAP_000.pdf